CLINICAL TRIAL: NCT01412060
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Cariprazine (RGH-188) in the Prevention of Relapse in Patients With Schizophrenia
Brief Title: A Study of Cariprazine in the Prevention of Relapse of Symptoms in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RGH-MD-06; 2011-002048-29 (EudraCT Number)
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic disorder
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There was no masking in the Open-Label Phase. There was masking in the Double-Blind Phase
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cariprazine - Open-label Phase (Experimental): Participants received 3, 6, or 9 mg cariprazine orally once a day for 6 weeks; the dose could be modified during this time. The cariprazine dose was fixed at 3, 6, or 9 mg for the last 14 weeks of this 20 week Open-label Phase.
  Interventions: Drug: Cariprazine
- Placebo - Double-blind Treatment Phase (Experimental): Participants received placebo orally once a day for 26 to 72 weeks.
  Interventions: Drug: Placebo
- Cariprazine - Double-blind Treatment Phase (Experimental): Participants received 3, 6, or 9 mg cariprazine orally once a day for 26 to 72 weeks
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Placebo — Placebo was supplied in capsules.
  Arms: Placebo - Double-blind Treatment Phase
Drug: Cariprazine — Cariprazine was supplied as 1.5 mg capsules (batch numbers BN0009242 and BN00018595) and 3 mg capsules.
  Other Names: RGH-188
  Arms: Cariprazine - Double-blind Treatment Phase; Cariprazine - Open-label Phase

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of cariprazine relative to placebo in the prevention of relapse of symptoms in participants with schizophrenia.

DETAILED DESCRIPTION:
There were 3 periods (phases) in the study. The Open-label Phase lasted 20 weeks. In the first 6 weeks, participants received 3, 6, or 9 mg cariprazine orally once a day; the dose could be modified during this time. The cariprazine dose was fixed at 3, 6, or 9 mg for the last 14 weeks of this Open-label Phase. At the end of Week 8, participants had to meet the following criteria to continue in the study.

* Positive and Negative Syndrome Scale (PANSS) total score ≤ 60 at the end of Week 8
* At least 20% decrease in PANSS total score from baseline to the end of Week 8
* Clinical Global Impressions - Severity (CGI-S) score ≤ 4 at the end of Week 8
* Score of ≤ 4 on each of the following 7 PANSS items: P1, P2, P3, P6, P7, G8, and G14 at the end of Week 8
* Stable dose during the previous 2 weeks
* No significant tolerability issues as judged by the Investigator at the end of Week 8

At the end of the Open-label Phase, participants were randomized into 2 treatment groups, cariprazine or placebo, if they met the following criteria:

* PANSS total score ≤ 60 at the end of Week 20
* At least 20% decrease in PANSS total score from baseline to the end of Week 20
* CGI-S score ≤ 4 at the end of Week 20
* Score of ≤ 4 on each of the following 7 PANSS items: P1, P2, P3, P6, P7, G8, and G14 at the end of Week 20
* No significant tolerability issues as judged by the Investigator During this Double-blind Treatment Phase, participants received either placebo or cariprazine at the same dosage (3, 6, or 9 mg) that they received during the last 14 weeks of the Open-label Phase.

All participants entered the 4 week Safety Follow-up Phase. They received a treatment other than the investigational product at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have provided informed consent prior to any study specific procedures.
* Participants currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) criteria for schizophrenia.
* Participants with normal physical examination, laboratory, vital signs, and/or electrocardiogram (ECG).
* Diagnosis of schizophrenia for a minimum of 1 year before Visit 1 (Screening).
* Positive and Negative Syndrome Scale (PANSS) total score ≥ to 70 and ≤ 120 at Visit 1 (Screening) and Visit 2 (beginning of Run-in Phase).
* Negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test (applies to female participants of childbearing potential only).
* Body mass index between 18 and 40 kg/m^2, inclusive.

Exclusion Criteria:

* Participants currently meeting DSM-IV-TR criteria for schizoaffective disorder, schizophreniform disorder, bipolar I and II and known or suspected borderline or antisocial personality disorder. or other DSM-IV-TR axis II disorders.
* Participants in their first episode of psychosis.
* Treatment-resistant schizophrenia over the last 2 years.
* Positive result from the blood alcohol test or from the urine drug screen for any prohibited medication.
* At imminent risk of injuring self or others or causing significant damage to property.
* Suicide risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 765 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2014-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, Study Director — Allergan
Locations (73):
- United States (25):
  - Forest Investigative Site 011, Little Rock, Arkansas
  - Forest Investigative Site 018, Cerritos, California
  - Forest Investigative Site 007, Costa Mesa, California
  - Forest Investigative Site 026, Culver City, California
  - Forest Investigative Site 008, Long Beach, California
  - Forest Investigative Site 002, Oceanside, California
  - Forest Investigative Site 019, Orange, California
  - Forest Investigative Site 001, Paramount, California
  - Forest Investigative Site 020, San Diego, California
  - Forest Investigative Site 005, Washington D.C., District of Columbia
  - Forest Investigative Site 024, Leesburg, Florida
  - Forest Investigative Site 017, Atlanta, Georgia
  - Forest Investigative Site 021, Chicago, Illinois
  - Forest Investigative Site 023, Baltimore, Maryland
  - Forest Investigative Site 010, Rockville, Maryland
  - Forest Investigative Site 003, Flowood, Mississippi
  - Forest Investigative Site 006, Creve Coeur, Missouri
  - Forest Investigative Site 014, St Louis, Missouri
  - Forest Investigative Site 012, Cedarhurst, New York
  - Forest Investigative Site 022, Dayton, Ohio
  - Forest Investigative Site 015, Austin, Texas
  - Forest Investigative Site 027, Austin, Texas
  - Forest Investigative Site 025, Dallas, Texas
  - Forest Investigative Site 013, Houston, Texas
  - Forest Investigative Site 009, Houston, Texas
- India (15):
  - Forest Investigative Site 305, Vijayawada, Andhra Pradesh
  - Forest Investigative Site 303, Ahmedabad, Gujarat
  - Forest Investigative Site 308, Ahmedabad, Gujarat
  - Forest Investigative Site 310, Ahmedabad, Gujarat
  - Forest Investigative Site 313, Mangalore, Karnataka
  - Forest Investigative Site 314, Manipal, Karnataka
  - Forest Investigative Site 301, Aurangabad, Maharashtra
  - Forest Investigative Site 306, Kalyān, Maharashtra
  - Forest Investigative Site 311, Nashik, Maharashtra
  - Forest Investigative Site 317, Jaipur, Rajasthan
  - Forest Investigative Site 302, Jaipur, Rajasthan
  - Forest Investigative Site 312, Madurai, Tamil Nadu
  - Forest Investigative Site 309, Kanpur, Uttar Pradesh
  - Forest Investigative Site 304, Lucknow, Uttar Pradesh
  - Forest Investigative Site 307, Varanasi, Uttar Pradesh
- Romania (12):
  - Forest Investigative Site 403, Bucharest
  - Forest Investigative Site 405, Bucharest
  - Forest Investigative Site 406, Bucharest
  - Forest Investigative Site 408, Bucharest
  - Forest Investigative Site 410, Bucharest
  - Forest Investigative Site 407, Campulung Muscel
  - Forest Investigative Site 412, Campulung Muscel
  - Forest Investigative Site 402, Constanța
  - Forest Investigative Site 411, Focşani
  - Forest Investigative Site 401, Iași
  - Forest Investigative Site 409, Iași
  - Forest Investigative Site 404, Târgovişte
- Slovakia (6):
  - Forest Investigative Site 508, Bratislava
  - Forest Investigative Site 507, Bratislava
  - Forest Investigative Site 504, Liptovský Mikuláš
  - Forest Investigative Site 505, Rimavská Sobota
  - Forest Investigative Site 503, Rožňava
  - Forest Investigative Site 506, Trnava
- Ukraine (15):
  - Forest Investigative Site 609, Kerch, AR Crimea
  - Forest Investigative Site 610, Dnipropetrovsk
  - Forest Investigative Site 613, Donetsk
  - Forest Investigative Site 616, Ivano-Frankivsk
  - Forest Investigative Site 605, Kharkiv
  - Forest Investigative Site 606, Kharkiv
  - Forest Investigative Site 604, Kharkiv
  - Forest Investigative Site 607, Kherson
  - Forest Investigative Site 602, Kyiv
  - Forest Investigative Site 601, Kyiv
  - Forest Investigative Site 612, Kyiv
  - Forest Investigative Site 603, Lviv
  - Forest Investigative Site 615, Odesa
  - Forest Investigative Site 611, Simferopol
  - Forest Investigative Site 608, Vinnytsia

REFERENCES:
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Correll CU, Potkin SG, Zhong Y, Harsanyi J, Szatmari B, Earley W. Long-Term Remission With Cariprazine Treatment in Patients With Schizophrenia: A Post Hoc Analysis of a Randomized, Double-Blind, Placebo-Controlled, Relapse Prevention Trial. J Clin Psychiatry. 2019 Jan 8;80(2):18m12495. doi: 10.4088/JCP.18m12495. PMID 30695290
- [Derived] Durgam S, Earley W, Li R, Li D, Lu K, Laszlovszky I, Fleischhacker WW, Nasrallah HA. Long-term cariprazine treatment for the prevention of relapse in patients with schizophrenia: A randomized, double-blind, placebo-controlled trial. Schizophr Res. 2016 Oct;176(2-3):264-271. doi: 10.1016/j.schres.2016.06.030. Epub 2016 Jul 15. PMID 27427558

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 765 participants were enrolled and received cariprazine in Run-in Phase; 751 of these, had at least 1 postbaseline Positive and Negative Syndrome Scale (PANSS) evaluation and 364 entered Stabilization Phase. Only 200 participants who completed Open-label phase, received either placebo (n=99) or cariprazine (n=101) in Double-Blind Phase.
Period: Open-label Run-in Period (RIP)
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase
Started | 765 | 0 | 0
Completed | 418 | 0 | 0
Not Completed | 347 | 0 | 0
Not completed — Adverse Event | 86 | 0 | 0
Not completed — Insufficient Therapeutic Response | 66 | 0 | 0
Not completed — Protocol Violation | 27 | 0 | 0
Not completed — Withdrawal of Consent | 117 | 0 | 0
Not completed — Lost to Follow-up | 32 | 0 | 0
Not completed — Other Miscellaneous Reasons | 19 | 0 | 0
Period: Period Between RIP and SP
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase
Started | 418 | 0 | 0
Completed | 364 | 0 | 0
Not Completed | 54 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Insufficient Therapeutic Response | 19 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Other Miscellaneous Reasons | 23 | 0 | 0
Period: Open-label Stabilization Period (SP)
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase
Started | 364 | 0 | 0
Completed | 264 | 0 | 0
Not Completed | 100 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0
Not completed — Insufficient Therapeutic Response | 9 | 0 | 0
Not completed — Protocol Violation | 14 | 0 | 0
Not completed — Withdrawal of Consent | 40 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0
Not completed — Other Miscellaneous Reasons | 19 | 0 | 0
Period: Period Between SP and DBP
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase
Started | 264 | 0 | 0
Completed | 200 | 0 | 0
Not Completed | 64 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal of Consent | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Did Not Met Criteria to Enter Next Phase | 4 | 0 | 0
Not completed — Other Miscellaneous Reasons | 55 | 0 | 0
Period: Double-blind Treatment Phase (DBP)
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase
Started | 0 | 99 | 101
Completed | 0 | 16 | 18
Not Completed | 0 | 83 | 83
Not completed — Adverse Event | 0 | 5 | 6
Not completed — Protocol Violation | 0 | 4 | 5
Not completed — Withdrawal of Consent | 0 | 10 | 15
Not completed — Lost to Follow-up | 0 | 6 | 5
Not completed — Other Miscellaneous Reasons | 0 | 11 | 27
Not completed — Relapse | 0 | 47 | 25

BASELINE CHARACTERISTICS:
Population: Run-in Phase safety population: All participants who received at least 1 dose of open-label cariprazine during the Run-in Phase of the study.
Arm/Group | Cariprazine - Open-label Phase
Number analyzed (Participants) | 765
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221
  Male | 544
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 728
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 149
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 313
  White | 299
  More than one race | 3
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 78.07 (20.10)
Height [Mean (Standard Deviation); unit: cm] | 170.98 (9.95)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.50 (5.63)
Waist circumference [Mean (Standard Deviation); unit: cm] | 90.39 (15.34)

OUTCOME MEASURES:

1. Primary Outcome: Time From Baseline to the First Symptom Relapse During the Double-blind Phase
Description: Relapse was defined as meeting ≥1 of the following criteria:1-Hospitalization due to worsening of condition;2-increase in Positive and Negative Syndrome Scale(PANSS) total score by ≥30% for participants,scored ≥50 or a ≥10-point increase for participants,scored <50 at randomization;3-increase in Clinical Global Impressions-Severity(CGI-S) score by ≥2 points at Week 20;4-deliberate self-injury or aggressive behaviour;5-suicidal/homicidal ideation judged clinically significant by Investigator;6-score of >4 on 1 or more of following PANSS items:P1,P2,P3,P6,P7,G8 or G14. Second assessment not performed based on Investigator discretion.
  PANSS is 30-item rating scale. Each item scored on 7-point scale. Total score ranges from 30 to 210. Lower score indicates fewer schizophrenic symptoms. CGI-S is 7-point scale,measures severity of participant's illness in comparison with others with same diagnosis. Lower score indicates less severe illness. 25th percentile for time to relapse was reported.
Time Frame: Up to 34 Weeks and Bi-Weekly thereafter until Week 92
Population: Double-blind intent-to-treat population: All participants who received at least 1 dose of double-blind investigational product and who had at least 1 post-randomization assessment of PANSS or CGI-S during the Double-blind Treatment Phase.
Measure: Number (95% Confidence Interval); unit: Days
Groups:
- Placebo: Participants received placebo orally once a day for 26 to 72 weeks. Placebo: Placebo was supplied in capsules.
- Cariprazine: Participants received 3, 6, or 9 mg cariprazine orally once a day for 26 to 72 weeks. Cariprazine: Cariprazine was supplied in capsules.
Arm/Group | Placebo | Cariprazine
Number analyzed (Participants) | 99 | 101
Days | 92 [44 to 151] | 224 [99 to NA] — The upper limit of the confidence interval could not be calculated due to insufficient number of events.
Statistical Analysis 1: Comparison: Placebo vs Cariprazine; Test type: Superiority or Other; p = 0.0010, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.28 to 0.73] — Hazard ratio (cariprazine 3-9 mg vs placebo) is based on Cox proportional hazards regression model, with treatment group as an explanatory variable

ADVERSE EVENTS:
Time Frame: First dose until 30 days after last dose of investigational product [Open-Label (Up to 184 days) and Double-Blind (Up to 536 days)]
Description: Run-in Phase Safety Population: All randomized participants who received at least 1 dose of investigational product and who had at least 1 post-randomization assessment of PANSS or CGI-S during the open-label phase (OLP) of the study.
  Double-blind Safety Population: All participants in the Randomized Population who took at least 1 dose of double-blind investigational product.
  Adverse events data was reported in periods as per the treatment received.
Groups:
- Open-label - Safety Follow-up Phase; Placebo - Safety Follow-up Phase; Cariprazine - Safety Follow-up Phase: Participants received no treatment during the 4 weeks Safety Follow-up Phase.
Arm/Group | Cariprazine - Open-label Phase | Placebo - Double-blind Treatment Phase | Cariprazine - Double-blind Treatment Phase | Open-label - Safety Follow-up Phase | Placebo - Safety Follow-up Phase | Cariprazine - Safety Follow-up Phase
All-Cause Mortality (participants affected / at risk) | 0/765 | 0/99 | 0/101 | 0/765 | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 50/765 | 14/99 | 14/101 | 6/765 | 2/99 | 0/101
Other Adverse Events (participants affected / at risk) | 425/765 | 28/99 | 35/101 | 0/765 | 0/99 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine - Open-label Phase (N=765) | Placebo - Double-blind Treatment Phase (N=99) | Cariprazine - Double-blind Treatment Phase (N=101) | Open-label - Safety Follow-up Phase (N=765) | Placebo - Safety Follow-up Phase (N=99) | Cariprazine - Safety Follow-up Phase (N=101)
Schizophrenia (Psychiatric disorders) | 19 | 7 | 5 | 3 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 10 | 2 | 2 | 3 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 5 | 0 | 0 | 0 | 0 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 3 | 0 | 2 | 0 | 0 | 0
Social stay hospitalisation (Social circumstances) | 2 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intentional product misuse (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Psychiatric evaluation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Psychotic behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Victim of crime (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine - Open-label Phase (N=765) | Placebo - Double-blind Treatment Phase (N=99) | Cariprazine - Double-blind Treatment Phase (N=101) | Open-label - Safety Follow-up Phase (N=765) | Placebo - Safety Follow-up Phase (N=99) | Cariprazine - Safety Follow-up Phase (N=101)
Constipation (Gastrointestinal disorders) | 39 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 46 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 48 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 49 | 0 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 148 | 0 | 0 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 55 | 3 | 6 | 0 | 0 | 0
Headache (Nervous system disorders) | 92 | 7 | 8 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 39 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 110 | 8 | 8 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 70 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 4 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 5 | 8 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 8 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 6 | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.